CLINICAL TRIAL: NCT04423432
Title: Effects of Creatine and Glucoseamine/ Chondritin Sulfate Co-Supplementation in Addition to Exercise and Physical Therapy in Patients With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Collaborators: Isra University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FUI/CTR/2020/4
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Electric Stimulation Therapy; Musculoskeletal Manipulations; Creatine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator)
  Interventions: Other: Lower Extremity Resistance Exercise Training; Other: Home Exercise Plan; Device: Electrotherapy + Heating; Procedure: Joint Mobilization
- Creatine Supplementation (Experimental)
  Interventions: Other: Lower Extremity Resistance Exercise Training; Other: Home Exercise Plan; Device: Electrotherapy + Heating; Procedure: Joint Mobilization; Dietary Supplement: Creatine Supplementation
- Glucoseamine/ Chondritin Sulfate Supplementation (Experimental)
  Interventions: Other: Lower Extremity Resistance Exercise Training; Other: Home Exercise Plan; Device: Electrotherapy + Heating; Procedure: Joint Mobilization; Dietary Supplement: Glucoseamine/ Chondritin Sulfate Supplementation

INTERVENTIONS:
Other: Lower Extremity Resistance Exercise Training — 3 times supervised exercise for 4 weeks Warm up (Self Paced walking for 10 minutes) leg press (8-12 RM) leg extension (8-12 RM) Sit to stand squat (with weight) Stationary Cycling (Maximum Resistance as per patient tolerance till failure)
  Other Names: Lower Extremity Strength Training
Other: Home Exercise Plan — 2 sets of 10 repetitions/day of
  1. AROM isolated knee extension and knee flexion
  2. Isometric isolated knee extension and knee flexion
  3. Isometric terminal knee extension
  4. Sit to stand squat
  terminal extension as Home Exercise Program (HEP). (Iwamoto J et al, 2007)
Device: Electrotherapy + Heating — Iinterferential Current therapy (2P), in combination with heating pad for 20 minutes
Procedure: Joint Mobilization — 1. Tibio-femoral Anterior Glide
  2. Tibio-femoral Posterior Glide
  3. Patellofemoral Joint Mobilization
  Other Names: Manual Therapy
Dietary Supplement: Creatine Supplementation — Creatine Supplementation 20g/day for 1 week followed by 5 g/day for 3 weeks
  Other Names: Creatine Monohydrate
  Arms: Creatine Supplementation
Dietary Supplement: Glucoseamine/ Chondritin Sulfate Supplementation — Glucoseamine/ Chondritin Sulfate Supplementation (500mg+400mg/day)
  Arms: Glucoseamine/ Chondritin Sulfate Supplementation

SUMMARY:
Osteoarthritis is the 11th highest contributor to disability world wide. In terms of conservative management of patients with knee osteoarthritis, Resistance exercise has been shown to be an effective intervention for reducing pain and cartilage degeneration and improving muscle strength, joint biomechanics and physical functioning. But, research shows that co supplementation can further augment the effects of resistance exercise. However, it is imperative to point out that the existing evidence is majorly focused on the individual effects of resistance exercise training and non-pharmacological supplementation, and is still deficient in the effects of co-supplementation in addition to resistance exercise training in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70 years
* Knee OA with history not less than three months.
* Radiological evidences of grade III or less on Kellgren classification.
* Knee pain on VNRS no more than 8/10

Exclusion Criteria:

* Neuromuscular conditions that may lead to fatigue such as multiple Sclerosis
* Signs of serious pathology (e.g., malignancy, inflammatory disorder, infection).
* History of trauma or fractures in lower extremity.
* Signs of lumbar radiculopathy or myelopathy.
* History of knee surgery or replacement.
* Patients on intra-articular steroid therapy within two months before the commencement of the study.
* Impaired skin sensation.
* Impaired renal function

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Knee Pain: Numeric Pain Rating Scale | 4 weeks
  Knee Pain will be quantified by using Numeric Pain Rating Scale
Knee Range of Motion | 4 weeks
  Knee Range of Motion will be quantified by using Gonimeter
Knee Isometric Muscle Strength | 4 weeks
  Knee Isometric Muscle Strength will be quantified by using Modified Sphygmomanometer Dynamometer
Six Minute Walk Test | 4 weeks
  Six Minute Walk Test will be used to quantify walking related performance fatigability, walkind distance and walking speed.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 4 weeks
  The KOOS is self-administered and assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life.
Body Composition | 4 weeks
  Body Composition will be quantified by using Bioelectrical Impedance
Fall Risk | 4 weeks
  Fall risk will be quantified by using Biodex balance System
Postural Stability | 4 weeks
  Postural Stability will be quantified by using Biodex balance System

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Osama, PhD*, Principal Investigator — Foundation University Institute of Rehabilitation Sciences
Locations (1):
- Foundation University Institute of Rehabilitation Sciences, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No